CLINICAL TRIAL: NCT06235892
Title: Prospective, Multicenter, Randomized, Open-label, Parallel-group Controlled Phase 3 Study of Tacrolimus Minimization in Kidney Transplant Recipients Selected According to the AGORA Algorithm for Their Low Immunological Risk and Medium-term Graft Failure
Brief Title: Tacrolimus Minimization in Kidney Transplant Recipients Selected According to the AGORA Algorithm for Their Low Immunological Risk and Medium-term Graft Failure
Acronym: AGORAC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC22_0525
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Organ Grafts
Keywords: Tacrolimus minimization; kidney transplant; AGORA Algorithm
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultra-low TACROLIMUS arm (Experimental): Ultra-low TACROLIMUS (TAC) arm based on MMF/MPA (Mycophenolate Mofetil/ Mycophénolic Acid) with or without CS (Cortico Steroid ) and TACROLIMUS to achieve 2-3.5 ng/ml trough levels during all the duration of the study.
  Interventions: Drug: TACROLIMUS
- SOC ( Standard of care)-TACROLIMUS arm (No Intervention): SOC-TAC arm based on MMF/MPA with or without CS and TACROLIMUS to achieve 4 and 7 ng/ml trough levels during all the duration of the study

INTERVENTIONS:
Drug: TACROLIMUS — TACROLIMUS 2-3.5 ng/ml
  Arms: Ultra-low TACROLIMUS arm

SUMMARY:
The goal of this clinical trial is that validation of the non-invasive biomarkers of the AGORA algorithm should make it possible to select patients with a very low immunological risk of graft failure to authorize safe minimization of their immunosuppression for adult patients at one-year post kidney transplantation.

The main question of the AGORAC trial is to demonstrate the impact of TACROLIMUS minimization using AGORA algorithm compared to standard of care on the kidney function 18 months after the minimization period.

ELIGIBILITY:
Inclusion Criteria:

* First kidney transplantation
* Living or brain death or
* Donation after circulatory death (Maastricht 3) donor,Compatible for ABO group with the donor,
* cPRA (Panel Reactive Antibody Calculated ) (or TGI: Incompatible Graft Rate )<20% on the day of the transplantation and no DSA (MFI <500) at pre transplant and at the time of the inclusion at one-year post transplantation (between 350 and 515 days after the transplantation.
* Eplet Mismatchs <= 14
* Normal or IFTA 1-2 histology on one-year surveillance biopsy.
* Patient insured under a health insurance scheme, according to national regulation.
* Patient (of childbearing age) with effective contraception.
* Patients treated with Tacrolimus (Prograf® or Advagraf®) and MMF / MPS (Mycophenolate Sodium) +/- Corticosteroid (CS)

Exclusion Criteria:

* Donation after circulatory death maastricht 2 (uncontrolled) and maastricht 1
* Pregnant women (serum or urine test), breastfeeding women
* Patient under legal protection (incl. under guardianship or trusteeship)
* Participation to a drug interventional study within 1 month prior to the inclusion
* Any retransplantation and combined transplantations and also other organ previous transplantations
* History of lymphoproliferative disorders
* Diagnosis of a malignant disease (according to the type of malignancy)
* Hepatitis C antibody or hepatitis B surface antigen (HbsAg) positive patient or HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Improvement of the renal function at 18 months after "ultra" minimization of Tacrolimus | Month 18
  Improvement will be assessed by measured glomerular filtration rate (mGFR) iohexol clearance.

SECONDARY OUTCOMES:
Incidence of biopsy-proven acute rejection (BPAR) according to the 2017 Banff classification (including borderline lesions) | Month 18
Type, severity and treatment of biopsy-proven acute rejection ( BPAR) | Month 18
Appearance of de novo donor-specific alloantibody (DSA) (4 digits and MFI treshold >500) | Month 18
Appearance or worsening of histological lesions of interstitial fibrosis and inflammatory tubular atrophy (IFTA) of study biopsy by considering that only patients with normal histology or with an IFTA-1 or 2will be randomized | Month 18
Prevalence of death, and graft loss (dialysis start or retransplantation) at end of study | Month 18
Prevalence of metabolic disorders: post-transplant diabetes mellitus (PTDM), dyslipidaemia and hypertension at end of study | Month 18
Treatment adherence consisting in monitoring immunosuppression adherence using Trackyourmed® to monitor individual variability tacrolimus intake | Month 18
Change in quality of life estimated using the EQ-5D ( EuroQol instrument - dimensions) questionnaire fulfilled by patients at baseline, Month 3, Month 6, Month 9, Month 12, Month15 and Month18 | Month 3, Month 6, Month 9, Month 12, Month15 and Month18
  There is two score in the EQ-5D-5L The first one is the descriptive system: Minimum value:5 ( no problems on any dimension) Maximum value: 25 ( extreme problems on all dimensions)
  The second score is EQ VAS (EuroQol vertical visual analogue scale) score. It is rated on a scale of 0-100 points. 0 points correspond to the worst possible health status, while 100 points correspond to the best possible health status.

CONTACTS AND LOCATIONS:
Locations (3):
- CHU de NANTES, Nantes, France
- Oslo University Hospital, Oslo, Norway
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No